CLINICAL TRIAL: NCT07279103
Title: The Effect of Multisensory Environment-Based Occupational Therapy Intervention on Sensory Processing, Cognitive, Behavioral Symptoms and Caregiver Burden in Alzheimer's Patients: A Randomized Controlled Study
Brief Title: Multisensory Environment-Based Occupational Therapy for Alzheimer's Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Medine Nur Özata Değerli, Research Assistant, Occupational Therapist, PhD Candidate, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9337fecbc0f54b90
Record Dates: First submitted 2025-11-19; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer s Disease; Occupational Therapy; Rehabilitation; Caregiver Burnout; Behavioral and Psychiatric Symptoms of Dementia; Sensory Processing Disorder; Cognitive
Keywords: Alzheimer's disease; dementia; occupational therapy; multisensory environment; sensory processing; cognitive function; behavioral and psychological symptoms; non-pharmacological intervention; caregiver burden
MeSH Terms: conditions — Caregiver Burden; Behavior; Alzheimer Disease; Dementia | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multisensory Environment-Based Occupational Therapy (Experimental): Participants in this arm will receive an exploratory, multisensory environment-based occupational therapy program.
  Interventions: Behavioral: Multisensory Environment-Based Occupational Therapy
- Occupational therapy (Experimental): Participants in this arm will receive a structured, directive occupational therapy program focusing on cognitive stimulation and daily living activities
  Interventions: Behavioral: Occupational therapy

INTERVENTIONS:
Behavioral: Multisensory Environment-Based Occupational Therapy — Participants will receive a multisensory environment-based occupational therapy intervention designed to expose them to structured sensory experiences. The intervention will last 4 weeks, delivered twice per week, for a total of 8 sessions, each lasting approximately 30 minutes. Sessions will be supportive and exploratory rather than directive.
  Before the intervention, each participant's sensory preferences, personal history, and cognitive status will be assessed to individualize the session content. Each session will follow a three-part structure consisting of preparation, main activity, and closing. During the main activity, the therapist will accompany the participant, facilitate engagement, and provide graded sensory options.
  The intervention will incorporate visual, auditory, tactile, proprioceptive, vestibular, olfactory, and taste stimuli. Examples include colored lighting, projected images, music, vibration tools, textured materials, movement-based activities, familiar scents
  Arms: Multisensory Environment-Based Occupational Therapy
Behavioral: Occupational therapy — The control group will not participate in any multisensory environment-based interventions. Instead, they will receive a directive occupational therapy program focused on cognitive stimulation and promoting independence in daily living activities. The intervention will last 4 weeks, with two sessions per week, totaling 8 sessions, each approximately 30 minutes.
  These sessions will not include purposeful multisensory experiences and will follow a structured, cognitively oriented approach tailored to the participant's abilities.
  Arms: Occupational therapy

SUMMARY:
This study aims to examine the effects of a multisensory environment-based occupational therapy intervention on sensory processing, cognitive status, behavioral and psychological symptoms, and caregiver burden in individuals diagnosed with Alzheimer's disease. Non-pharmacological approaches in Alzheimer's management have been shown to slow functional decline, reduce behavioral symptoms, and improve caregivers' well-being. Multisensory environments provide visual, auditory, tactile, proprioceptive, vestibular, olfactory, and gustatory stimuli to support sensory integration and enhance engagement, particularly in individuals with cognitive and communication difficulties. The study will be conducted using a randomized controlled design and will include individuals aged 65 years and older with moderate-stage Alzheimer's disease and their primary caregivers. The intervention will be implemented over four weeks with two sessions per week. Outcome measures will include the Adult/Adolescent Sensory Profile,Loewenstein Occupational Therapy Cognitive Assessment-Geriatric version, Neuropsychiatric Inventory, and Zarit Caregiver Burden Inventory. The study is expected to contribute to the evidence base supporting sensory-based occupational therapy interventions in dementia care.

DETAILED DESCRIPTION:
This study aims to investigate the effects of a multisensory environment-based occupational therapy intervention on sensory processing, cognitive functions, behavioral and psychological symptoms, and caregiver burden in individuals diagnosed with Alzheimer's disease. Alzheimer's disease, as a progressive neurodegenerative condition, leads to gradual impairments in cognitive, emotional, and functional abilities, which in turn cause behavioral disturbances and significantly increase caregiver stress. In recent years, non-pharmacological approaches have gained attention for their role in managing dementia-related symptoms, maintaining daily functioning, and supporting caregivers' well-being.

Multisensory environments, which offer structured stimulation involving visual, auditory, tactile, proprioceptive, vestibular, olfactory, and gustatory senses, are designed to facilitate sensory integration and promote engagement through meaningful sensory experiences. These environments can reduce agitation, enhance communication, and improve mood and attention among individuals with dementia by creating a sense of comfort and familiarity.

This randomized controlled study will include individuals aged 65 years and older who have been clinically diagnosed with moderate-stage Alzheimer's disease, as well as their primary caregivers. The intervention will be implemented over a four-week period, consisting of two 45-minute sessions per week conducted in a controlled multisensory therapy room. Standard care will be provided to the control group.

Outcome measures will include the Adult/Adolescent Sensory Profile to assess sensory processing patterns, the Lowenstein Occupational Therapy Cognitive Assessment for Geriatrics version for cognitive performance, the Neuropsychiatric Inventory for behavioral and psychological symptoms, and the Zarit Caregiver Burden Inventory for caregiver stress. Pre- and post-intervention assessments will be conducted to determine changes in the target variables.

It is anticipated that the multisensory environment-based occupational therapy intervention will positively affect sensory processing and cognitive functions, reduce behavioral and psychological symptoms, and alleviate caregiver burden. The findings of this study are expected to provide strong empirical support for the integration of sensory-based occupational therapy interventions into dementia care programs, contributing to both clinical practice and the growing body of evidence on non-pharmacological rehabilitation approaches for Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria

Age 65 years or older

Clinical diagnosis of Alzheimer-type dementia according to DSM-5 criteria

Moderate stage dementia:

Global Deterioration Scale Stage 5

Mini-Mental State Examination score between 10 and 18

Living at home with a primary caregiver

Presence of a primary caregiver who can accompany the participant during therapy sessions

Basic literacy level (ability to read and write at a minimal functional level)

Application to or referral from the Occupational Therapy Departments of Çankırı Karatekin University or Hacettepe University

Exclusion Criteria

Presence of additional chronic, neurological, or sensory problems that impair communication

e.g., uncorrected visual impairment

e.g., uncorrected hearing impairment

Prior receipt of any non-pharmacological therapy specifically targeting dementia

Any medical or psychiatric condition that may interfere with participation or assessments

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive Status | 8 week
  The Loewenstein Occupational Therapy Cognitive Assessment-Geriatric Version is a cognitive assessment battery used by occupational therapists to identify cognitive impairments that affect daily functioning and quality of life in older adults. The tool includes a structured assessment kit, a manual, and scoring guidelines. It evaluates six cognitive domains-orientation, perception, praxis, visuomotor organization, thinking operations, and memory-through 23 subtests. The assessment kit contains various materials such as colored blocks, tangrams, grooming items, sequencing cards, picture booklets, categorization cards, a pegboard, and a clock-drawing sheet. The manual provides instructions on administering the subtests and scoring each item. Scores range from 1 to 4 depending on performance. Therapists conduct the assessment using the standardized materials and record the results on the scoring form. It is a commercially available assessment and is accessible in
Sensory Processing | 8 week
  Adult Sensory Profile (ASP):
  The Adult Sensory Profile was developed to evaluate sensory response patterns related to sensory systems in adults. Based on Ayres' Sensory Integration Theory, the profile aims to assess behavioral response patterns that indicate sensory processing difficulties across specific sensory systems, including over-responsivity, under-responsivity, and sensory seeking. Over-responsivity refers to heightened reactions to ordinary stimuli that typically do not bother others; under-responsivity refers to a lack of awareness of stimuli that most people would notice; and sensory seeking refers to behaviors characterized by actively pursuing sensory input with higher intensity or frequency than usual. The ASP consists of 11 factors and 48 items, scored on a 5-point Likert scale (1: never, 2: rarely, 3: sometimes, 4: often, 5: always). The Turkish validity and reliability study of the scale has also been conducted.
Behavioral and Psycological symptoms | 8 week
  Neuropsychiatric Inventory:
  This inventory will be used to assess behavioral and psychological symptoms associated with dementia. Developed in 1994, it evaluates delusions, hallucinations, agitation, depression, anxiety, euphoria, apathy, disinhibition, irritability, abnormal motor behaviors, sleep/nighttime problems, and changes in appetite/eating habits. Each subdomain is rated based on frequency (0-4), severity (0-3), and caregiver distress (0-5). Subdomain scores are calculated by multiplying frequency and severity. The total inventory score is obtained by summing all subdomain scores. The minimum possible score is 0 and the maximum is 144. Scores between 0-20 indicate mild symptoms, 21-50 indicate moderate symptoms, and scores above 50 indicate severe behavioral and psychological symptoms related to dementia. The Turkish validity and reliability study of the inventory reported a Cronbach's alpha value of 0.79.
Caregiver burden | 8 week
  Caregiver Burden Inventory:
  This inventory was developed to measure the impact of caregiving. It consists of 24 items rated on a 0-4 Likert scale and includes five subscales: (a) time-dependence burden, (b) developmental burden, (c) physical burden, (d) social burden, and (e) emotional burden. The total score ranges from 0 to 100, with higher scores indicating a greater level of caregiver burden. The Turkish validity and reliability study reported high internal consistency, with Cronbach's alpha values of 0.94 for the total scale and similarly high reliability coefficients for each subscale.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe Universitesi, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and the sensitive nature of dementia-related clinical information.

REFERENCES:
- [Result] Ravn MB, Klingberg T, Petersen KS. The Adult Sensory Profile in Care Homes Targeting People Diagnosed with Dementia: A Qualitative Study from the Care Provider Perspective. Rehabil Res Pract. 2018 Aug 5;2018:5091643. doi: 10.1155/2018/5091643. eCollection 2018. PMID 30155306
- [Result] Berthiaume, K., Craig, B., & Rayford, B. S. (2024). The collaboration between occupational therapy and psychology in treating adolescents in a psychiatric residential treatment facility. Multisensory immersion room as a treatment intervention. Occupational Therapy in Mental Health, 40(2), 123-137.
- [Result] Bennett S, Laver K, Voigt-Radloff S, Letts L, Clemson L, Graff M, Wiseman J, Gitlin L. Occupational therapy for people with dementia and their family carers provided at home: a systematic review and meta-analysis. BMJ Open. 2019 Nov 11;9(11):e026308. doi: 10.1136/bmjopen-2018-026308. PMID 31719067
- [Result] Baker R, Holloway J, Holtkamp CC, Larsson A, Hartman LC, Pearce R, Scherman B, Johansson S, Thomas PW, Wareing LA, Owens M. Effects of multi-sensory stimulation for people with dementia. J Adv Nurs. 2003 Sep;43(5):465-77. doi: 10.1046/j.1365-2648.2003.02744.x. PMID 12919265
- [Result] Baker R, Bell S, Baker E, Gibson S, Holloway J, Pearce R, Dowling Z, Thomas P, Assey J, Wareing LA. A randomized controlled trial of the effects of multi-sensory stimulation (MSS) for people with dementia. Br J Clin Psychol. 2001 Mar;40(1):81-96. doi: 10.1348/014466501163508. PMID 11317951
- [Result] Ayres, A. J. (1972). Sensory integration and learning disorders. (No Title).
- [Result] Akça Kalem Ş, H. H., Cummings JL, Gürvit H. (2005). Validation study of the Turkish translation of the Neuropsychiatric Inventory. 21st International Conference of Alzheimer's Disease International, İstanbul, Turkey.